CLINICAL TRIAL: NCT00348478
Title: Determination of the Impact of Water and Health Education on Trachoma and Ocular C. Trachomatis in Niger
Brief Title: Impact of Water and Health Education Programs on Trachoma and Ocular C. Trachomatis in Niger
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: World Vision (Other); CONRAD (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA00001455
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2005-11

CONDITIONS: Trachoma
Keywords: trachoma; chlamydia trachomatis; water; health education; face washing
MeSH Terms: conditions — Trachoma; Health Education | interventions — Water

INTERVENTIONS:
Behavioral: water and health education program to improve hygiene

SUMMARY:
There are no specific trials addressing the benefit of water provision and health education on prevalence of trachoma and infection with ocular Chlamydia trachomatis over time, despite considerable effort to provide water resources in trachoma endemic areas. Such information is sorely needed, to advance the Global Alliance agenda for the Elimination of Blinding Trachoma. This community-based clinical trial will randomize ten communities in Maradi Niger, half to receive delivery of water and health education services, and half for delivery of services at a later date. We hypothesize that the intervention communities will have lower rates of trachoma and C. trachomatis one and two years after delivery of services compared to communities without such services. This trial will provide, for the first time, solid evidence of the effect of such services on trachoma, as well as the added benefit following antibiotic provision by the Ministry of Health on sustaining reductions in trachoma and infection.

DETAILED DESCRIPTION:
Objectives

This study has the following objectives:

1. To determine the effect on clinical trachoma in a cohort of children from baseline to one, two, and three years post-intervention with a village-based water and health education program.
2. To determine the effect on ocular C. trachomatis infection in a cohort of children from baseline to one, two, and three years post-intervention with a village-based water and health education program.
3. A secondary outcome is the measure of under five years mortality in intervention compared to control

Study Design:

Population: We are proposing to evaluate trachoma over time in a sample of children age 1-5 years at baseline in villages in Niger where World Vision is planning immediate water and health education services delivery, compared to a sample of children in villages where services will be implemented after two years.

Services: World Vision plans water wells to serve a population of about 300, in villages of about 300-5,000 persons. Thus each village has around 1-17 wells. The goal is to provide water within 500 meters with a wait time of less than 15 minutes. Health education on use of water and hygiene practices is also part of services delivery. A World Vision Area Development Program officer establishes and trains a water and sanitation committee to provide health education for their village. Villages who are randomly selected to be part of these services will be classified as "intervention" villages. In addition, there are other villages where the planning process has just started and wells would not be drilled for over two years. Villages who are randomly selected to be in the group where services will not be available immediately, will be classified as "control" villages.

Design:

Overview The design is a three-year longitudinal study of trachoma and infection with ocular Chlamydia trachomatis in a cohort of children age 1-5 at baseline. From a list of villages in Maradi region that are intended to have a water program within the next three years, we will randomly select six villages to be the "intervention" villages and six villages to be the "control" villages. We will aim to include 360 children, randomly selected from the 6 "intervention" villages (one per mother for a total of up to 60 in each village) and 360 children randomly selected from 6 "control" villages. Surveys for trachoma and infection will be carried out at baseline, one, two, and three years from baseline. Details are described below.

Villages The 1995 census of Maradi was the basis for selecting villages in the Kornaka West district of Maradi, Niger, where World Vision is planning their intervention. The villages in the study should be of comparable size (between 900-2,100 [estimated] persons), as village size may be an important predictor of trachoma status at 12 months.

The villages were selected as follows:

1. A list of all villages with an estimated population between 900 and 2,100 in the district of Kornaka West was generated. The total number of villages was 18
2. The Area Development Program (ADP) geographic area was stratified so that control villages would not be within 5 KM of villages where there was a village with a well.
3. Each village was assigned a sequential number from a table of random numbers. The six villages with the lowest numbers assigned in the "left" strata were selected as the "intervention" villages, and the six villages with the lowest numbers in the "right" strata were selected as the "control" villages. Four additional villages with the next lowest numbers were selected as reserve villages, in case they are needed because a village refuses to have the survey.

This selection process means that World Vision will plan to work first in the six villages designated as "intervention villages", so they have wells and health education programs within the first year. World Vision will not implement water and health education programs in the "control" villages until after two years. The rest of the villages not selected as either intervention or controls can have programs implemented as decided by World Vision to suit their needs with the understanding that wells will not be implemented in villages within 5 KM of control villages until after two years. The reserve villages will be released if not needed as soon as the census is completed.

Census

Once the villages have been selected, a team of trained census-takers will do three things: gather minimal data on the village, minimal data on each compound or "concession", and do a complete census of everyone in the concession. Every concession must have a census to provide an accurate count of the number of persons and number of children age 1-5 years old.

The senior census taker will do the following:

* Explain the study to the village leadership so that they understand what is being asked of the village residents.
* Explain that children in the survey sample found to have trachoma will be treated with topical tetracycline during the surveys. However, not every child in every household is part of the survey and antibiotics are restricted to just these survey children. However, mass treatment for these communities where everyone is treated is planned by the government at the end of two years.
* Secure permission of the village leadership to conduct the village survey, concession survey, and trachoma survey on a sample of children age 1-5 years.
* Collect the village information
* Identify persons in the village who can lead the census team to all concessions in the village for the information on the concession and the census.
* Supervise the team of census takers to carry out the census of the village.
* Certify that all households/concessions in the village have a census form at the end of the village census

The census takers will be responsible for collecting the concession information and the complete census on every concession/household in the village.

* Collect the data on each concession from the chef of the concession, and by observation, on the "Questionniare Chef du Concession"
* Collect information on everyone in the

Selection of Sample of Children

Once the census of all concessions is completed, the random sample of up to 60 children age 1 to 5 years and 5 months in each village can be selected. A stratified random sampling strategy will be developed that limits the selection to no more than one children per mother, with preference for 0 to 1 child age 1 to 5 and 5/12 months for a total of 60 per village. This strategy minimizes clustering of children within households, which is possible if a simple random sample is used.

Survey for Trachoma

Baseline surveys for trachoma in the sample of children age 1-5 5/12 years will take place prior to any water or health education intervention.

The surveys will consist of the following steps:

1. Prior to the survey in the village, a member of the team will alert the village leadership that the survey team is coming, which households are in the survey, and to make sure that the sample children stay in the village for the days of the survey.
2. The day of the survey, the mothers will be asked to bring their sample children to a survey site close by, for the examination. As they come, consent will be obtained by the senior trachoma grader, and the name will be checked on the list, and a form and a single specimen label filled out for the examiner and the laboratory technician.
3. The trachoma grader will be everting the eyelids. He must change gloves between each child, even children in the same house, and even if the child does not appear to have trachoma. The trachoma grader, wearing 2.5X loupes, will assess the trachoma status of the tarsal plate, using the WHO Simplified grading scheme.
4. While the left eyelid is still everted, the laboratory technician, following careful procedures described in the training manual, will roll the swab three times across the tarsal plate to obtain a specimen.
5. If the child has TF or TI, the mother is given a tube of tetracycline and instructions on proper use for that child.
6. At the end of each day in the field, all specimens are transferred to a freezer in World Vision in Maradi, awaiting return to the freezer in Niamey. During the drive to Niamey, specimens must be kept frozen as well, with ice packs.

By 6 months into the first year, the water and health education program in the "intervention" villages should be underway, and the well completed. This assures at least 6 months exposure to the intervention before the next survey at one year.

The same sample of children will be surveyed for trachoma at one, two, and three years. No additional children will be added to the sample to replace any who have died or moved away. The procedures for the follow up surveys are exactly the same as for the baseline survey.

Mass Treatment will be provided by the Ministry of health after the Second Year Survey; control villages will receive water and sanitation programs at that time.

The "intervention villages" continue with water and sanitation, and undergo mass treatment after two year survey. The "control villages, where implementation of water and health education are planned for implementation after the second year survey, also receive mass treatment of azithromycin. For the third year, we can compare the prevalence of trachoma after three years of water and health education plus mass treatment, to mass treatment plus shorter exposure to water and health education.

At the same time as the other surveys, the complete census list of all children age five and under will be updated for new children added , and children who were deceased in the previous year. These data will be used to determine the under five mortality for the villages in the previous year. A comparison of under five years mortality for the intervention and control villages will be done at the end of the three year surveys.

Comparison of trachoma and ocular C. trachomatis infection in sentinel children resident in intervention villages compared to sentinel children resident in control villages at one and two years post baseline will be done. A secondary comparison is to determine the under five years mortality at two and three years post baseline in intervention versus control villages.

ELIGIBILITY:
Inclusion Criteria:

* villages size between 900-2100 residents as of 1995 census in Kornaka West district of Niger
* village leadership approval of entry of village in the study
* sentinel children ages 6 months to 5 years and five months

Exclusion Criteria:

* village already has health education program for hygiene
* village within 5 km of a well
* child already has a sibling in the study population

Ages: 6 Months to 65 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720
Dates: Start 2005-12; Study Completion 2008-01

PRIMARY OUTCOMES:
trachoma
ocular C. trachomatis infection

SECONDARY OUTCOMES:
under five years mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K West, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States